CLINICAL TRIAL: NCT00833703
Title: Long Term Safety Study in Patients Included in the CLARINET Study With Cyanotic Congenital Heart Disease Palliated With a Systemic-to-pulmonary Artery Shunt and for Whom the Shunt is Still in Place at One Year of Age
Brief Title: Long Term Safety of Clopidogrel in Neonates/Infants With Systemic to Pulmonary Artery Shunt Palliation
Acronym: CLARINET LT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTS10916; 2008-004999-53 (EudraCT Number)
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2011-08-16 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Heart Defects, Congenital
Keywords: cyanotic congenital heart disease; shunt palliation; thrombosis; clopidogrel
MeSH Terms: conditions — Heart Defects, Congenital; Thrombosis | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 0.2 mL/kg/day matching placebo solution once daily.
  Interventions: Drug: placebo
- Clopidogrel 0.2 mg/kg/day (Experimental): 0.2 mL/kg/day Clopidogrel reconstituted solution at 1mg/mL once daily.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Form: reconstituted solution using Clopidogrel powder
  Route: oral or enteric
  Frequency: once daily
  Dose: daily dose adjusted for weight
  Other Names: SR25990; Plavix
  Arms: Clopidogrel 0.2 mg/kg/day
Drug: placebo — Form: reconstituted solution using matching placebo powder
  Route: oral or enteric
  Frequency: once daily
  Dose: daily dose adjusted for weight
  Arms: Placebo

SUMMARY:
This study is the extension of the CLARINET study [NCT00396877 -EFC5314] in neonates or infants with cyanotic congenital heart disease palliated with a systemic-to-pulmonary artery shunt.

The primary objective was to assess the safety up to 18 months of age of the extended use of Clopidogrel 0.2 mg/kg/day in patients for whom the shunt was still in place at one year of age.

The secondary objective was to assess the efficacy on the occurrence of shunt thrombosis requiring intervention or any death.

DETAILED DESCRIPTION:
Patients remained in the treatment group to which they were originally allocated for the CLARINET study and continued blindly their treatment (0.2 mg/kg/day of clopidogrel or placebo) up to the occurrence of shunt thrombosis, next surgical procedure for correction of the congenital heart disease, death, or 18 months of age, whichever came first. The maximum treatment duration were 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients randomized in the CLARINET study,
* Still receiving the study drug,
* Palliative systemic-to-pulmonary artery shunt still in place at 1 year of age,
* Investigator's decision to continue based on his/her judgment of the expected benefit / risk of continuing treatment with study drug,
* Signed informed consent to participate in the long-term safety study.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (15):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Derived] Avlonitis VS, Planas S, Hayes AM, Parry A. Occlusion of modified Blalock-Taussig shunt after clopidogrel cessation. Ann Thorac Surg. 2012 Feb;93(2):656-8. doi: 10.1016/j.athoracsur.2011.07.071. PMID 22269735

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 participants were enrolled between January 2009 and January 2010 in 25 sites in 15 countries (7 countries involved in CLARINET study were not selected as the delay in obtaining IRB/IEC and Health Authorities approvals would prevent recruitment and/or no patient would be recruited as the second surgery is always performed before 1 year of age).
Period: Overall Study
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day
Started | 23 (Included) | 26 (Included)
Treated | 23 | 26
Completed Treatment | 22 | 24
Completed | 23 (Completed follow-up) | 25 (Completed follow-up)
Not Completed | 0 | 1
Not completed — Parent(s)/guardian(s)'s request | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day | Total
Number analyzed (Participants) | 23 | 26 | 49
Age Continuous [Mean (Standard Deviation); unit: days]
  at randomization in CLARINET study | 45.2 (26.1) | 33.1 (20.5) | 38.8 (23.8)
  at inclusion | 368.1 (4.2) | 368.0 (2.7) | 368.0 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  United States | 0 | 1 | 1
  Portugal | 3 | 1 | 4
  Taiwan | 4 | 5 | 9
  Spain | 0 | 2 | 2
  Russian Federation | 1 | 0 | 1
  United Kingdom | 1 | 2 | 3
  Italy | 0 | 1 | 1
  India | 0 | 1 | 1
  France | 0 | 1 | 1
  Hungary | 2 | 1 | 3
  Mexico | 6 | 4 | 10
  Brazil | 4 | 2 | 6
  Malaysia | 1 | 1 | 2
  Poland | 1 | 1 | 2
  Germany | 0 | 3 | 3
Weight at inclusion [Mean (Standard Deviation); unit: kilograms (kg)] | 7.9 (1.1) | 8.1 (1.2) | 8.0 (1.2)
Height at inclusion [Mean (Standard Deviation); unit: centimeters (cm)] | 71.8 (2.8) | 70.0 (10.4) | 70.8 (7.8)
Type of initial shunt palliation [Number; unit: participants]
  Modified Blalock Taussig Shunt with Norwood | 0 | 1 | 1
  Modified Blalock Taussig Shunt without Norwood | 18 | 20 | 38
  Sano procedure with Norwood | 0 | 0 | 0
  Sano procedure without Norwood | 1 | 1 | 2
  Central shunt | 1 | 3 | 4
  Stent of ductus arteriosus | 3 | 1 | 4
Shunt on cardiopulmonary bypass [Number; unit: participants]
  Yes | 2 | 5 | 7
  No | 21 | 21 | 42
Age at shunt palliation [Mean (Standard Deviation); unit: days] | 25.7 (28.7) | 13.7 (12.7) | 19.4 (22.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bleeding Events
Description: All bleeding events experienced during the study period were collected as for any Adverse Event.
  The 'on-treatment' period was defined as the period from inclusion in the extension study up to 28 days after treatment discontinuation, and participants who experienced bleeding events during that period were counted.
Time Frame: Up to a maximum of 6 months
Population: The analysis was performed on the Intent-to-treat (ITT) population that consisted of all included participants. Participants were analyzed in the treatment arm allocated at randomization into the CLARINET study.
Measure: Number; unit: participants
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day
Number analyzed (Participants) | 23 | 26
participants
  Any bleeding event | 0 | 2
  - Serious | 0 | 0
  - Serious with an outcome of death | 0 | 0
  - Leading to permanent treatment discontinuation | 0 | 0

2. Secondary Outcome: Number of Participants With Shunt Thrombosis Requiring Intervention or Deaths
Description: Outcome events, shunt thrombosis requiring intervention or death, experienced during the study period were recorded.
  Participants were counted excluding the events that occured after the participant's protocol study end (occurrence of shunt thrombosis, next surgical procedure for correction of the congenital heart disease, death, or 18 months of age, whichever came first).
Time Frame: Up to a maximum of 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day
Number analyzed (Participants) | 23 | 26
participants
  shunt thrombosis requiring intervention | 0 | 0
  death | 1 | 0

3. Primary Outcome: Number of Participants According to Bleeding Type/Etiology
Description: For all reported bleeding events, the type and the etiology of the bleeding event were collected. Participants who experienced bleeding events during the 'on-treatment period' were counted by bleeding type and etiology.
Time Frame: Up to a maximum of 6 months
Population: The analysis was performed on the same population as previously (i.e. ITT population).
Measure: Number; unit: participants
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day
Number analyzed (Participants) | 23 | 26
participants
  Spontaneous | 0 | 1
  Puncture (vascular access site) | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to a maximum of 6 months. All Adverse Events (AE) experienced during the study period were collected regardless of seriousness or relationship to the drug .
Description: The analysis was performed on the intent-to-treat population and included all AE that developed/worsened during the 'on-treatment period' (i.e. from inclusion in the extension study up to 28 days after treatment discontinuation).
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 3/23 | 6/26
Other Adverse Events (participants affected / at risk) | 7/23 | 17/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Clopidogrel 0.2 mg/kg/Day (N=26)
Bronchiolitis (Infections and infestations) | 0 | 1
Croup infectious (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Low cardiac output syndrome (Cardiac disorders) | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=23) | Clopidogrel 0.2 mg/kg/Day (N=26)
Any infections and infestations (Infections and infestations) | 6 | 14
Upper respiratory tract infection (Infections and infestations) | 0 | 6
Gastroenteritis (Infections and infestations) | 2 | 2
Ear infection (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 0 | 2
Pharyngitis (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Any gastrointestinal disorders (Gastrointestinal disorders) | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Any general disorders and administration site conditions (General disorders) | 1 | 6
Pyrexia (General disorders) | 0 | 4
Any respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Any injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 | 3
Any skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 | 2
Any cardiac disorders (Cardiac disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can publish the results. Prior to publication, the sponsor shall review the manuscript and can request changes, provided they do not jeopardize the accuracy and/or the scientific value of the publication. The approval is given in writing by the sponsor, not exceeding 90 days.